CLINICAL TRIAL: NCT00261144
Title: Collagenase in the Treatment of Cellulite
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Marie A. Badalamente, Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Cell 101
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite | interventions — Collagenases; Biological Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Collagenase — One 0.58mg injection every two weeks for six weeks (total three 0.58mg injections)
Biological: Biological — Collagenase injection
  Other Names: Collagenase

SUMMARY:
The purpose of this study is to determine if collagenase injection will reduce or eliminate the appearance of cellulite of the thigh.

DETAILED DESCRIPTION:
This is an open label study of collagenase injection therapy for reduction and/or elimination of cellulite of the posterolateral thighs.

ELIGIBILITY:
Inclusion Criteria:

* 10 x 10 cm area of cellulite of the posterolateral thigh(s)

Exclusion Criteria:

* any chronic, serious or uncontrolled medical condition
* inability to conform to study visits (12-15 per year)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Reduction and/or elimination of cellulite in the posterolateral thigh | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Badalamente, PhD, Principal Investigator — Dept. Orthopaedics, SUNY@Stony Brook, NY 11794; Alexander B Dagum, MD, Principal Investigator — Dept. Surgery, SUNY@Stony Brook, NY 11794
Locations (1):
- Dept. Orthopaedics, SUNY Stony Brook, Stony Brook, New York, United States